CLINICAL TRIAL: NCT02227758
Title: Peripheral Nerve Stimulation Registry for Intractable Migraine Headache
Acronym: Relief
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: NM-11-059-EU-ON
Record Dates: First submitted 2014-04-16; First posted 2014-08-28 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Intractable Chronic Migraine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- implanted chronic migraine patients: Patients diagnosed with chronic migraine, failed 3 or more preventative drugs, with at least moderate disability, and implanted with a St. Jude Medical Conformité Européenne approved implantable neurostimulation system

SUMMARY:
The purpose of this study is to evaluate the long-term safety and performance of neurostimulation for the treatment of intractable chronic migraine as well as to detect infrequent complications or problems only apparent in "real-world" practice

ELIGIBILITY:
* Patient is 18 years of age or older.
* Patient has signed and received a copy of the Informed Consent form;
* Patient has been implanted with a St. Jude Medical CE approved implantable neurostimulation system for the treatment of intractable chronic migraine:

  * Patient diagnosed with chronic migraine (15 or more days per month with headache lasting at least 4 hours per day)
  * Patient has failed three or more preventative drugs for treatment of their migraine
  * Patient has at least moderate disability determined using a validated migraine disability instrument [e.g., MIDAS >11 or HIT-6 >56]

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with intractable chronic migraine and implanted with a St.Jude Medical conformité européenne approved implantable neurostimulation system
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Belgium (2):
  - Heilig Hartziekenhuis, Roeselare, West-Vlaanderen
  - Centre Hospitalier Régional de la CITADELLE, Liège
- Germany (7):
  - Klinikum Delmenhorst GmbH, Delmenhorst, Großherzogtum Oldenburg
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Praxis fur Neurologie, Spezielle Schmerztherapie, Psychotherapie, Essen, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Migräne and Kopfschmerzklinik Königstein, Königstein, Saxony
  - Schmerzklinik und Praxis an der Schmerzklinik Kiel, Kiel, Schleswig-Holstein
  - Neurologische Klinik und Poliklinik Charité Campus Mitte, Berlin
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Spain (3):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario, Madrid
  - Hospital Puerta de Hierro, Madrid
- Karolinska Hospital, Stockholm, Stockholm County, Sweden
- United Kingdom (4):
  - John Radcliffe hospital, Oxford, Oxfordshire
  - Royal London Hospital, London, Royal London Hospital
  - Seacroft Hospital, Leeds, Yorkshire
  - King's College Hospital, London

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Implanted Chronic Migraine Patients
Started | 112
Completed | 45
Not Completed | 67

BASELINE CHARACTERISTICS:
Arm/Group | Implanted Chronic Migraine Patients
Number analyzed (Participants) | 112
Age, Continuous [Mean (Full Range); unit: years] | 45.9 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 33
Region of Enrollment [Number; unit: participants]
  Sweden | 1
  Belgium | 3
  Luxembourg | 1
  United Kingdom | 18
  Germany | 83
  Spain | 6

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (First 12 Weeks)
Description: Events were classified as hardware related when a malfunction or migration of any device component including leads, extensions, IPG's, occurred. Events will classified as biological in cases where there was a biological reaction (hematoma, pain, etc.) to either the device or the surgical procedure to implant the device. Events were classified as stimulation related if the event was known to be caused by stimulation.
Time Frame: 3 months
Measure: Number; unit: events
Arm/Group | Implanted Chronic Migraine Patients
Number analyzed (Participants) | 112
events
  Hardware-related AE | 17
  Biological AE | 27
  Stimulation related AE | 5
  Other AE | 1

2. Primary Outcome: Headache Pain Relief
Description: Patient reported headache pain relief in percentage for the previous month; patients were asked about their pain relief in percentage in the previous month; patient were asked "in the last month", how much headache relief has the implant provided (0% represents no relief, 100% represents complete relief)
Time Frame: 3 months
Population: 82 patients had available data for pain relief in the previous month at the 3 month follow-up visit
Measure: Mean (Full Range); unit: percentage pain relief
Arm/Group | Implanted Chronic Migraine Patients
Number analyzed (Participants) | 82
percentage pain relief | 25.1 [0 to 100]

3. Primary Outcome: Headache Days
Description: Percentage change in number of Headache days from Baseline to 3 Months. Headache days are the amount of days the subject had an headache in the previous 3 months as captured by the MIDAS questionnaire.
Time Frame: 3 months
Population: 69 patients had available data for headache days in the previous 3 months at the 3 month follow-up visit
Measure: Mean (Standard Deviation); unit: percent change in headache days
Arm/Group | Implanted Chronic Migraine Patients
Number analyzed (Participants) | 69
percent change in headache days | -16 (0.71)

4. Primary Outcome: Migraine Disability
Description: Percentage change in Midas score from Baseline to 3 Months. The Midas questionnaire consists out of 5 questions to be answered by the patient. Three questions address the number of missed days due to headache in school or paid work, household work and family, social or leasure activities. The two remaining questions document the number of additional days with significant limitations to activity (defined as at least 50% reduced productivity) in the domains of employment and household work. The total score is the sum of days completed for questions 1-5. Midas score ranges from 0 to 21+ with higher values indicating greater disability.
Time Frame: 3 months
Population: 63 patients had available data for all 5 questions of the Midas questionnaire computing the total score at the 3 month follow-up visit. Excluding the outliers, 59 patients had available data.
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Midas Score Including 4 Outliers: Including outliers with a reported increase of 128%, 148%, 225% and 434% at 3 months.
- Midas Score Excluding 4 Outliers: Excluding outliers with a reported increase of 128%,148%, 225%, 434%
Arm/Group | Midas Score Including 4 Outliers | Midas Score Excluding 4 Outliers
Number analyzed (Participants) | 63 | 59
percentage of change | 74 (6.2) | -37 (0.4)

5. Primary Outcome: Patient Satisfaction
Description: Patients very satisfied or satisfied with the headache relief since the implant. Patients were asked about their satisfaction (very satisfied, satisfied, neither satisfied or dissatisfied, unsatisfied, very unsatisfied)
Time Frame: 3 months
Population: 84 subjects had available data for patient satisfaction at the 3 month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Chronic Migraine Patients
Number analyzed (Participants) | 84
Participants | 28

6. Primary Outcome: Physician Satisfaction
Description: Patients for who the physician is very satisfied or satisfied with the patient headache relief since the implant. Physicians were asked about their satisfaction (very satisfied, satisfied, neither satisfied or dissatisfied, unsatisfied, very unsatisfied)
Time Frame: 3 months
Population: 84 subjects had available data for physician satisfaction at the 3 month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Chronic Migraine Patients
Number analyzed (Participants) | 84
Participants | 43

7. Primary Outcome: Quality of Life
Description: Patients who reported the change in overall quality of life since the implant with greatly improved or improved. Patients were asked about their change in overall quality of life (Greatly improved, improved, neither improved or deteriorated, deteriorated, greatly deteriorated)
Time Frame: 3 months
Population: 83 subjects had available data for Quality of life at the 3 month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Chronic Migraine Patients
Number analyzed (Participants) | 83
Participants | 32

8. Primary Outcome: Quality of Life
Description: Patients for who the physician reported the change in overall quality of life of the patient since the implant with greatly improved or improved. Physicians were asked about the change in overall quality of life of the patient(Greatly improved, improved, neither improved or deteriorated, deteriorated, greatly deteriorated)
Time Frame: 3 months
Population: 84 subjects had available data for physician reported overall quality of life
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Chronic Migraine Patients
Number analyzed (Participants) | 84
Participants | 43

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Serious Device Related Adverse Events are described. The AE's reported on clinicaltrials.gov have a threshold of 5%
Groups:
- Implanted Chronic Migraine Patients: Patients diagnosed with chronic migraine, failed 3 or more preventative drugs, with at least moderate disability, and implanted with a St. Jude Medical Conformité Européenne approved implantable neurostimulation system who experienced a Serious Device related adverse event
Arm/Group | Implanted Chronic Migraine Patients
Serious Adverse Events (participants affected / at risk) | 26/112
Other Adverse Events (participants affected / at risk) | 7/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted Chronic Migraine Patients (N=112)
Breakage/facture of the extension (Product Issues) | 2 (2)
Device Malfunction (Product Issues) | 2 (2)
IPG migration (Skin and subcutaneous tissue disorders) | 2 (2)
Infection: IPG and lead site (Infections and infestations) | 2 (2)
Infection: lead site only (Infections and infestations) | 3 (3)
Lead breakage/fracture (Product Issues) | 2 (2)
Lead migration (Skin and subcutaneous tissue disorders) | 8 (8)
persistant pain and/or numbness: IPG site only (Skin and subcutaneous tissue disorders) | 1 (1)
persistant pain and/or numbness: lead site only (Skin and subcutaneous tissue disorders) | 1 (1)
persistent pain at connector site (Skin and subcutaneous tissue disorders) | 1 (1)
skin erosion (Skin and subcutaneous tissue disorders) | 2 (2)
Wound site complications (Skin and subcutaneous tissue disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted Chronic Migraine Patients (N=112)
Persistent pain and/or numbness (Surgical and medical procedures) | 7 (7) — For 7 patients, there were reports of persistent pain and/or numbness at the lead and/or IPG site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less